CLINICAL TRIAL: NCT07320092
Title: Comparison of the Incidence of Atelectasis Assessed by Lung Ultrasound in Patients Undergoing Surgery in Supine and Prone Positions
Brief Title: Supine vs Prone Position and Atelectasis Assessed by Lung Ultrasound
Acronym: LUS-ATELEC
Status: Recruiting | Type: Observational
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, CHINARA NAMAZOVA, Research Assistant, Istanbul University - Cerrahpasa
Other Study IDs: E-74555795-050.04-1231752; 2025/24 (Other: Istanbul University-Cerrahpasa)
Record Dates: First submitted 2025-12-22; First posted 2026-01-06 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Postoperative Atelectasis
Keywords: Lung Ultrasound; Atelectasis; Supine Position; Prone Position; General Anesthesia; Perioperative Care
MeSH Terms: conditions — Pulmonary Atelectasis; Deception

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Supine Position: Patients undergoing surgery in the supine position under general anesthesia.
- Prone Position: Patients undergoing surgery in the prone position under general anesthesia.

SUMMARY:
Atelectasis frequently develops during and after general anesthesia due to factors such as anesthesia-induced diaphragmatic dysfunction, reduced functional residual capacity, altered ventilation-perfusion matching, and surgical positioning. The development of atelectasis has been associated with postoperative hypoxemia and other pulmonary complications.

Lung ultrasound (LUS) has emerged as a reliable, radiation-free bedside imaging modality for the detection and monitoring of atelectasis. LUS allows assessment of lung aeration through standardized ultrasound patterns and scoring systems, enabling dynamic evaluation in the perioperative period.

This is a prospective, observational cohort study designed to compare the incidence and severity of atelectasis in patients undergoing surgery in the supine position versus the prone position under general anesthesia. Adult patients undergoing elective surgical procedures will be enrolled. No experimental intervention will be applied, and all anesthetic and surgical management will follow routine clinical practice.

Lung ultrasound examinations will be performed at predefined time points after induction of anesthesia and before extubation. A standardized lung ultrasound protocol and scoring system will be used to assess lung aeration loss and detect the presence of atelectasis.

The primary outcome of the study is the difference in atelectasis detected by lung ultrasound between supine and prone surgical positions. The secondary outcome is the change in lung ultrasound scores over time.

This study aims to clarify the effects of supine and prone positions on perioperative atelectasis and to support the clinical use of lung ultrasound as a noninvasive monitoring tool in perioperative and anesthetic practice..

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18 years or older.
* Patients scheduled for elective surgery under general anesthesia.
* Patients undergoing surgery in the supine or prone position.
* Patients able to provide informed consent.

Exclusion Criteria:

* Emergency surgical procedures.
* Pre-existing severe pulmonary disease affecting lung ultrasound assessment.
* Hemodynamic instability requiring urgent intervention.
* Contraindications to lung ultrasound examination.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients aged 18 years and older who are scheduled to undergo elective surgical procedures under general anesthesia. Patients will be evaluated according to surgical positioning (supine or prone) during routine perioperative care.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-09-15 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Difference in lung ultrasound-detected atelectasis between supine and prone surgical positions | Perioperative (After induction of general anesthesia and before extubation)
  Lung aeration will be evaluated using the Lung Ultrasound Score (LUS), a semiquantitative scoring system assessing aeration loss in 12 lung regions.
  In the supine position, lung ultrasound assessment will be performed along:
  the parasternal line (intercostal spaces 1-4 and 4-8), the anterior axillary line (intercostal spaces 1-6 and 6-12), and the posterior axillary line (intercostal spaces 1-6 and 6-12).
  In the prone position, lung ultrasound assessment will be performed along:
  the paravertebral line (intercostal spaces 1-6 and 6-12), the posterior axillary line (intercostal spaces 1-6 and 6-12), and the anterior axillary line (intercostal spaces 1-6 and 6-12). Each lung region will be scored from 0 to 3, resulting in a total LUS ranging from 0 to 36, where higher scores indicate greater loss of aeration and more severe atelectasis.
  Assessments will be performed after induction of general anesthesia and before extubation.

CONTACTS AND LOCATIONS:
Overall Officials: ÖZLEM KORKMAZ DİLMEN, PROFESSOR, Principal Investigator — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University-Cerrahpasa, Cerrahpasa Faculty of Medicine, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared, as this is a single-center observational study conducted for a postgraduate thesis.

REFERENCES:
- [Background] Bouhemad B, Brisson H, Le-Guen M, Arbelot C, Lu Q, Rouby JJ. Bedside ultrasound assessment of positive end-expiratory pressure-induced lung recruitment. Am J Respir Crit Care Med. 2011 Feb 1;183(3):341-7. doi: 10.1164/rccm.201003-0369OC. Epub 2010 Sep 17. PMID 20851923
- [Background] Tusman G, Böhm SH, Warner DO, Sprung J. Atelectasis and perioperative pulmonary complications in general anesthesia. Br J Anaesth. 2012;108(2):229-240. PMID: 22156255.
- [Background] Acosta CM, Maidana GA, Jacovitti D, Belaunzaran A, Cereceda S, Rae E, Molina A, Gonorazky S, Bohm SH, Tusman G. Accuracy of transthoracic lung ultrasound for diagnosing anesthesia-induced atelectasis in children. Anesthesiology. 2014 Jun;120(6):1370-9. doi: 10.1097/ALN.0000000000000231. PMID 24662376
- [Background] Monastesse A, Girard F, Massicotte N, Chartrand-Lefebvre C, Girard M. Lung Ultrasonography for the Assessment of Perioperative Atelectasis: A Pilot Feasibility Study. Anesth Analg. 2017 Feb;124(2):494-504. doi: 10.1213/ANE.0000000000001603. PMID 27669555
- [Background] Lichtenstein DA. Lung ultrasound in the critically ill. Ann Intensive Care. 2014 Jan 9;4(1):1. doi: 10.1186/2110-5820-4-1. PMID 24401163